CLINICAL TRIAL: NCT05951478
Title: Primary Ciliary Dyskinesias: Identification of Specific Severity Criteria and Phenotype-genotype Correlation Study
Brief Title: DCP (RaDiCo Cohort) (RaDiCo-DCP)
Acronym: DCP
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-74
Record Dates: First submitted 2022-05-06; First posted 2023-07-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Ciliary Dyskinesias (PCD) are rare, autosomal recessive respiratory diseases, due to a defect in mucociliary clearance linked to abnormalities in the structure and/or function of the cilia. The variety of ciliary abnormalities identified reflects the genetic heterogeneity of PCDs. The thirty or so genes currently implicated explain the pathology in about half of the patients. PCDs are characterized by recurrent infections of the upper (rhinosinusitis) and lower (bronchitis) airways, beginning in early childhood and progressing respectively to nasal polyposis and bronchial dilatation. In half of the cases, there is a lateralization defect of the organs (situs inversus) corresponding to Kartagener's syndrome. There is more frequent infertility in men (immobility of spermatozoa) than in women (miscarriages and tubal pregnancies). About a third of patients progress to respiratory failure. The identification of predictive factors of severity, specific to PCDs, would improve patient care. It is also important to assess the quality of life of patients with PCD, particularly at the ENT level.

Data from prevalent patients are currently integrated into three separate and complementary databases: the "e-RespiRare" database, the "DCP Cils" database and the "DCP genes" database. The first step is therefore to constitute the RaDiCo-DCP database which will include data from prevalent and incident patients whose diagnosis of PCD is certain.

The cohort aims to improve the routine care of PCD patients, in particular by highlighting predictive factors of severity, allowing early and personalized care, to assess the social impact (quality of life) and medical conditions of ENT impairment, as well as adult infertility, to finely characterize the ciliary phenotype. The study also aims to search for new DCP genes and to allow genotype/phenotype correlation studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient fulfilling at least one of the following criteria for PCD confirmed diagnosis: Kartagener's syndrome and/or specific anomaly of the ciliary ultrastructure and/or an unambiguous mutation in a PCD gene
* Having at least one annual follow-up visit

Non-inclusion Criteria:

* Patients with an unconfirmed diagnosis of PCD
* Patients with an evolving concomitant pathology that may interfere with the assessment of PCD-related manifestations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes children and adults with the confirmed diagnosis of PCD. The objective is to recruit 300 patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison and description for severe and non-severe patients of the phenotypic characteristics of the disease in adult and pediatric patients. | Through study completion, an average of 5 years

SECONDARY OUTCOMES:
Validation of the involvement of new DCP genes | Through study completion, an average of 5 years
  Validation of the involvement of new DCP genes highlighted in the context of medical care will be done by association study in well-defined subgroups of patients.
Impact of disease on quality of life will be evaluated through scores of quality of life questionnaires Best Cilia 6-12 years old | Through study completion, an average of 5 years
Impact of disease on quality of life will be evaluated through scores of quality of life questionnaire Best Cilia 13-17 years old | Through study completion, an average of 5 years
Impact of disease on quality of life will be evaluated through scores of quality of life questionnaire Best Cilia 18+ years old | Through study completion, an average of 5 years
Impact of disease on quality of life will be evaluated through scores of quality of life questionnaire Sino-nasal outcome test-22 | Through study completion, an average of 5 years

OTHER OUTCOMES:
Association studies between the different clinical phenotypic aspects, the ciliary phenotype and the genotype. | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard MAITRE, Principal Investigator — INSERM UMR 955
Locations (28):
- France (28):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Pellegrin-Enfants, Bordeaux
  - CHU de Caen, Caen
  - Hôpital Clémenceau, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital Le Bocage, Dijon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Femme-Mère-Enfant, Lyon
  - Hôpital Louis Pradel, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Lenval, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Tenon, Paris
  - American Memorial Hospital, Reims
  - Hôpital Charles Nicolle, Rouen
  - Hospices Civils, Strasbourg
  - Hôpital Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Hôpital Larrey, Toulouse
  - Hôpital de Clocheville, Tours